CLINICAL TRIAL: NCT06328933
Title: A Randomized Controlled Trial to Explore the Effect of Intermittent Oro-esophageal Tube on Feeding Amount
Brief Title: Intermittent Oral Tube on Feeding Amount
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copka Sonpashan (Other Government)
Responsible Party: Sponsor-Investigator, Copka Sonpashan, The Research Director, Chao Phya Abhaibhubejhr Hospital
Organization: Chao Phya Abhaibhubejhr Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IOE feeding amount
Record Dates: First submitted 2024-03-10; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Oro-esophageal Tube Feeding+comprehensive rehabilitation therapy (Experimental): Assigned randomly before the treatment, all patients were provided with comprehensive rehabilitation therapy as follows:
  Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
  The observation group was given enteral nutritional support with Intermittent Oro-esophageal Tube according to the following procedure. The feeding content was formulated by the nutritionists based on the condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups
  Interventions: Device: Intermittent Oro-esophageal Tube Feeding; Behavioral: comprehensive rehabilitation therapy
- Nasogastric Tube Feeding+comprehensive rehabilitation therapy (Active Comparator): Assigned randomly before the treatment, all patients were provided with comprehensive rehabilitation therapy as follows:
  Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
  Besides, the control group was given enteral nutritional support with Nasogastric Tube according to the relevant guidelines. Within 4 hours after admission, the placement of the feeding tube was conducted by professional medical staffs and after intubation, the tube was secured to the cheek with medical tape. The feeding was conducted once every 3-4 hours, with 200-300ml each time. The total feeding volume was determined based on daily requirements.
  Interventions: Device: Nasogastric Tube Feeding; Behavioral: comprehensive rehabilitation therapy

INTERVENTIONS:
Device: Nasogastric Tube Feeding — The control group was given enteral nutritional support with Nasogastric Tube Feeding according to the relevant guidelines. Within 4 hours after admission, the placement of the feeding tube was conducted by professional medical staffs and after intubation, the tube was secured to the patient's cheek with medical tape. The feeding was conducted once every 3-4 hours, with 200-300ml each time. The total feeding volume was determined based on daily requirements. The feeding content was formulated by the nutritionists based on the patients condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups. For patients with limited tube feeding compliance, we made appropriate adjustments to ensure that they were not at risk of severe malnutrition as much as possible.
  Arms: Nasogastric Tube Feeding+comprehensive rehabilitation therapy
Device: Intermittent Oro-esophageal Tube Feeding — The observation group was given enteral nutritional support with Intermittent Oro-esophageal Tube according to the following procedure: Before each feeding, inside and outside of the tube was cleaned with water. During feeding, the patient should maintain a semi-reclining or sitting position with mouth opened, and the tube was inserted slowly and smoothly into the upper part of the esophagus by medical staffs while the appropriate depth of intubation was checked with the calibration markings on the tube wall. The distance from the incisors to the head part of the tube should be between 22-25 cm. However, the specific depth should be evaluated based on patients' feedback and adjusted accordingly. After insertion, the tail part of the tube should be put into a container full of water and the absence of continuous bubbles indicated a successful intubation. Then, the feeding was to be conducted three times per day with 50 ml per minute and 400-600ml for each feeding.
  Arms: Intermittent Oro-esophageal Tube Feeding+comprehensive rehabilitation therapy
Behavioral: comprehensive rehabilitation therapy — Including： Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.

SUMMARY:
The goal of this clinical trial is to compare the differences in feeding amount and nutritional status between ischemic stroke patients using Intermittent Oro-esophageal Tube and Nasogastric Tube. Patients will be randomly divided into an observation group and a control group, all receiving routine rehabilitation treatment. On this basis, the observation group will use Intermittent Oro esophageal Tube for enteral nutrition support, while the control group will use Nasogastric Tube. Researchers will compare changes in daily intake and nutritional status of two groups of patients before and after the study to see if Intermittent Oro-esophageal Tube can improve the feeding amount and nutritional status between ischemic stroke patients compared to Nasogastric Tube

DETAILED DESCRIPTION:
The study will last 15 days for each participant. The goal of this clinical trial is to compare the differences in feeding amount and nutritional status between ischemic stroke patients using Intermittent Oro-esophageal Tube and Nasogastric Tube. Patients will be randomly divided into an observation group and a control group, all receiving routine rehabilitation treatment. On this basis, the observation group will use Intermittent Oro esophageal Tube for enteral nutrition support, while the control group will use Nasogastric Tube. Researchers will compare changes in daily intake and nutritional status of two groups of patients before and after the study to see if Intermittent Oro-esophageal Tube can improve the feeding amount and nutritional status between ischemic stroke patients compared to Nasogastric Tube

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* Meeting the diagnostic criteria for ischemic stroke .
* Dysphagia confirmed by Videofluoroscopic Swallowing Study.
* Clear consciousness.
* No history of prior stroke.
* Stable vital signs.

Exclusion Criteria:

* Dysphagia that might be caused by other diseases that might cause dysphagia, such as head and neck tumors, traumatic brain injury, myasthenia gravis, etc.
* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Simultaneously in need to undergo other therapy that might affect the outcomes of this study.
* Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Nutritional status-total protein | day 1 and day 15
  The relevant indicators include total protein (TP, g/L) from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach ones and in the morning.
Nutritional status-hemoglobin | day 1 and day 15
  The relevant indicators include hemoglobin (Hb, g/L)from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach ones and in the morning.
Nutritional status-albumin | day 1 and day 15
  The relevant indicators include albumin (ALB, g/L)from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach ones and in the morning.
Nutritional status-prealbumin | day 1 and day 15
  The relevant indicators include prealbumin (PA, mg/L) from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach ones and in the morning.

SECONDARY OUTCOMES:
Feeding Amount | day 1 and day 15
  The total amount of nutrients consumed by the patient on the day was recorded, excluding fresh water, units: milliliters
Body weight | day 1 and day 15
  Body weight measurement of the infants was conducted by the same nurse according to the relevant standards.
Functional Oral Intake Scale | day 1 and day 15
  During Dysphagia-Functional Oral Intake Scale assessment, evaluators engage in communication with the patient, conduct observations, and make records to assess the patient's oral intake ability. The Functional Oral Intake Scale assessment form includes seven levels of scoring, ranging from level 1 to level 7, indicating a progressive improvement in the patient's oral intake ability. In general, the result below level 6 indicates unsafe for oral intake while level 6 and above indicates that eating via mouth can be safely conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Li, Study Chair — Site Coordinator of United Medical Group located in Miami